CLINICAL TRIAL: NCT03410108
Title: A Single-Arm, Multicenter, Phase 2 Study of Brigatinib in Japanese Patients With ALK-Positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase 2 Study of Brigatinib in Japanese Participants With Anaplastic Lymphoma Kinase (ALK)-Positive Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brigatinib-2001; U1111-1204-8752 (Other: WHO); JapicCTI-183823 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2022-06

CONDITIONS: ALK-positive Advanced NSCLC
Keywords: Drug therapy
MeSH Terms: interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brigatinib 90 mg + Brigatinib 180 mg (Experimental): Brigatinib 90 milligram (mg), tablets, orally, once daily (QD) for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onward cycles of 28 days until investigator-assessed progressive disease (PD) or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to Cycle 34 of 28-day cycle, until data cut-off date 29 September 2020.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablet

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of brigatinib in Japanese participants with anaplastic lymphoma kinase (ALK)-positive NSCLC.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib. Brigatinib is being tested in participants with ALK-positive NSCLC in order to evaluate efficacy and safety of oral doses of brigatinib in Japanese participants with ALK-positive NSCLC.

The study will enroll approximately 110 participants. Participants will be enrolled in non-randomized and opened manner:

- Brigatinib 90 mg for the first 7 days, followed by Brigatinib 180 mg of Brigatinib tablets, once daily in a 28-days cycle.

All participants will be asked to take tablets of brigatinib once daily with or without food throughout the study.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 53 months. Participants will make multiple visits to the clinic during the treatment period, and posttreatment period including a follow-up assessment after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Japanese participants aged >=20 years on the day of consent.
2. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
3. Have histologically or cytologically confirmed stage IIIB, stage IIIC (locally advanced or recurrent and not a candidate for definitive multimodality therapy), or stage IV NSCLC.
4. Have documentation of ALK rearrangement that meets following criteria.

   For the Safety Evaluation Lead-in Part and the Refractory Expansion Part, participants must meet 1 of the following 2 criteria:
   1. Have documentation of ALK rearrangement by a positive result from the Vysis ALK Break Apart fluorescence in situ hybridization (FISH) Probe Kit, the Nichirei Histofine ALK iAEP Kit, or the Ventana ALK (D5F3) Companion Diagnostics (CDx) Assay at any time during prior disease course. The sponsor may require an adequate tissue available for central laboratory testing by the Vysis ALK Break Apart FISH test if a documented ALK rearrangement is confirmed by a positive result from the Nichirei Histofine ALK iAEP Kit "ONLY".
   2. Had a documented ALK rearrangement by a different test at any time during prior disease course, and adequate tissue available for central laboratory testing by the Vysis ALK Break Apart FISH test. Central confirmation of ALK rearrangement is not required before enrollment.

   For TKI-naïve Expansion Cohort, participants must meet the following criteria Have documentation of ALK rearrangement by a positive result from Ministry of Health, Labour and Welfare (MHLW) Approved tests (e.g Vysis ALK Break Apart FISH Probe Kit, the Nichirei Histofine ALK iAEP Kit, or the Ventana ALK [D5F3] CDx Assay) prior to enrollment, and required to submit sufficient tumor tissue for central laboratory testing upon request of sponsor. Central confirmation of ALK rearrangement is not required before enrollment
5. The Refractory Expansion Part only: had documented progressive disease (PD) during treatment or within 30 days after discontinuation of treatment with ALK inhibitor.

   * Note 1: The Refractory Expansion Part consists of the Main Cohort and a Sub-cohort based on prior ALK inhibitor treatment. The Main Cohort includes participants who had previously received alectinib (as their only ALK inhibitor) or both crizotinib and alectinib (regardless the sequence of those 2 ALK inhibitors), and a total of 47 participants will be enrolled. Participants with all other sequences of up to 2 prior ALK inhibitor(s) may be included in the Sub-cohort, and the number of participants will be limited to 20.
   * Note 2: Participants who will be included in the Main Cohort of the refractory should have documented PD during treatment or within 30 days after discontinuation of treatment with alectinib.
6. Have at least 1 measurable (ie, target) lesion per RECIST version 1.1. Note: Previously irradiated lesions may not be used for target lesions, unless there is unambiguous radiological progression after radiotherapy. Brain lesions may not be used as target lesions if they were 1) previously treated with whole brain radiation therapy (WBRT) within 3 months, or 2) previously treated by stereotactic radiosurgery (SRS) or surgical resection.
7. Recovered from toxicities related to prior anticancer therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 Grade =<1. Note: Treatment-related alopecia is allowed.
8. Have a life expectancy of >=3 months.
9. Have adequate organ and hematologic function, as determined by:

   1. Both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =<2.5 times the upper limit of the normal range (ULN) (=<5×ULN is acceptable if liver metastases are present).
   2. Total serum bilirubin =<1.5×ULN (<3.0×ULN for participants with Gilbert syndrome).
   3. Serum creatinine <1.5×ULN. For participants with creatinine levels above or equal to 1.5×ULN, the participant is eligible if the estimated creatinine clearance using the Cockcroft-Gault formula is >=30 mL/minute.
   4. Serum lipase =<1.5×ULN and serum amylase =<1.5×ULN.
   5. Absolute neutrophil count (ANC) >=1.5×10^9/Liter (L).
   6. Platelet count >=75×10^9/L.
   7. Hemoglobin >=9 gram (g)/ deciliter (dL).
   8. Percutaneous oxygen saturation (SpO2) >=94% without oxygen support. Participants who need oxygen support are excluded.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of =<2.
11. Must meet the following criteria:

    1. Female participants who:

       * Are postmenopausal for at least 1 year before the screening visit, OR
       * Are surgically sterile, OR
       * If they are of childbearing potential, agree to practice 1 highly effective non-hormonal method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, OR
       * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant, from the time of signing the informed consent through 4 months after that last dose of study drug. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
    2. Male participants, even if surgically sterilized (ie, status postvasectomy), who:

       * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, OR
       * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant, during the entire study treatment period and through 4 months after that last dose of study drug. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
12. Have the willingness and ability to comply with scheduled visit and study procedures.

Exclusion Criteria:

1. Previously received the following treatments. The Refractory Expansion Part only: received any prior ALK inhibitor not specified in the protocol.

   TKI-naïve Expansion Cohort only: received any prior TKI including but not limited to ALK inhibitor and vascular endothelial growth factor receptor (VEGFR) TKI.
2. The Refractory Expansion Part only: received more than 2 prior ALK inhibitors. Note: The Safety Evaluation Lead-in Part allows participants with any line of prior ALK inhibitor which includes treatment-naïve participants; however, ALK inhibitor-naïve participants may be enrolled after the confirmation of first 3 dose-limiting toxicity (DLT) evaluable participants to have no more than 1 DLT during Cycle 1 by investigator's judgement.
3. The Safety Evaluation Lead-in Part and the Refractory Expansion Part only: received ALK inhibitor within 7 days before the first dose of brigatinib.
4. Previously received more than 1 regimen (more than 3 regimens in the Safety Evaluation Lead-in part) of systemic anticancer therapy (other than ALK inhibitors) for locally advanced or metastatic disease. Note: A systemic anticancer therapy regimen will be counted if it is administered over at least 1 cycle. A new anticancer agent used as maintenance therapy will be counted as a new regimen unless it was previously used as initial anticancer therapy. Neoadjuvant or adjuvant systemic anticancer therapy will be counted as a prior regimen if completion of (neo) adjuvant therapy occurred <12 months before the first dose of brigatinib.
5. Treatment with any investigational products within 30 days or 5 half-lives of that investigational agent, whichever is longer, before the first dose of brigatinib.
6. Received chemotherapy or radiation within 14 days before the first dose of brigatinib, except stereotactic radiosurgery (SRS) or stereotactic body radiation therapy.
7. Received antineoplastic monoclonal antibodies within 30 days before the first dose of brigatinib.
8. Received systemic treatment with strong inhibitors or strong and moderate inducers of cytochrome P450 (CYP) 3A within 7 days before the first dose of brigatinib.
9. Had major surgery within 30 days before the first dose of brigatinib. Minor surgical procedures such as venous catheter placement or minimally invasive biopsies are allowed.
10. Have been diagnosed with another primary malignancy other than NSCLC, except for the following adequately/definitively treated malignancies: nonmelanoma skin cancer, cervical cancer in situ, nonmetastatic prostate cancer; or participant with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
11. Have symptomatic central nervous system (CNS) metastases (parenchymal or leptomeningeal) at screening or asymptomatic disease requiring an increasing dose of corticosteroids to control symptoms within 7 days before the first dose of brigatinib. Note: If a participant has worsening neurological symptoms or signs due to CNS metastasis, the participant needs to complete local therapy and be neurologically stable (with no requirement for an increasing dose of corticosteroids or use of anticonvulsants for symptomatic control) for 7 days before the first dose of brigatinib.
12. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Participants with asymptomatic leptomeningeal disease and without cord compression are allowed.
13. Have ongoing or history of interstitial lung disease (ILD) (including interstitial pneumonitis, pneumonitis, radiation pneumonitis, drug-related pneumonitis, organized pneumonia, and pulmonary alveolitis).
14. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not limited to:

    1. Myocardial infarction within 6 months before the first dose of brigatinib.
    2. Unstable angina within 6 months before the first dose of brigatinib.
    3. Congestive heart failure within 6 months before the first dose of brigatinib.
    4. Uncontrolled atrial arrhythmias despite appropriate medical therapy.
    5. History of ventricular arrhythmia, including history of ventricular tachycardia, ventricular fibrillation, or torsades de pointes. Participants with premature ventricular contractions are allowed.
    6. Cerebrovascular accident or transient ischemic attack within 6 months before the first dose of brigatinib.
15. Have uncontrolled hypertension. Participants with hypertension should be under treatment at the start of screening and demonstrate adequate control of blood pressure.
16. Have an ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics.
17. Have a known history of human immunodeficiency virus (HIV) infection. Testing is not required in the absence of history.
18. Hepatitis B surface antigen (HBsAg) positive, detectable hepatitis B viral load, or detectable hepatitis C virus (HCV) infection viral load. Note: Participants who have positive hepatitis B core antibody (HBcAb) or hepatitis B surface antibody (HBsAb) can be enrolled but must have an undetectable hepatitis B viral load. Participants who have positive HCV antibody can be enrolled but must have an undetectable hepatitis C viral load.
19. Have malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of brigatinib.
20. Have a known or suspected hypersensitivity to brigatinib or its excipients.
21. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period. Note: Female participants who are lactating will be excluded, even if they discontinue breastfeeding.
22. Have any condition or illness that, in the opinion of the investigator, would compromise participant safety or interfere with the evaluation of brigatinib.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- Japan (33):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Matsuzaka Citizen's Hospital, Matsuzaka, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Cancer Center, Shinden, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mok T, Nishio M, Yoshida T, Ahn MJ, Kudou K, Asato T, Yang H, Tong X, Vincent S, Zhang P, Yamamoto N, Kim ES. Efficacy and safety of brigatinib after alectinib in patients with ALK-positive NSCLC: Integrated analysis of the ALTA-2 and J-ALTA studies. Lung Cancer. 2025 Nov;209:108793. doi: 10.1016/j.lungcan.2025.108793. Epub 2025 Oct 9. PMID 41110382
- [Derived] Sugawara S, Kondo M, Yokoyama T, Kumagai T, Nishio M, Goto K, Nakagawa K, Seto T, Yamamoto N, Kudou K, Asato T, Zhang P, Ohe Y. Brigatinib in Japanese patients with tyrosine kinase inhibitor-naive ALK-positive non-small cell lung cancer: first results from the phase 2 J-ALTA study. Int J Clin Oncol. 2022 Dec;27(12):1828-1838. doi: 10.1007/s10147-022-02232-7. Epub 2022 Aug 29. PMID 36036294
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b601c4db2bf003ab493a8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with non-small cell lung cancer (NSCLC) based on prior anaplastic lymphoma kinase-tyrosine kinase inhibitor (ALK-TKI) treatment or naïve (with no prior treatment with TKIs) took part in the study at 32 investigative sites in Japan from 29 January 2018 to data cut-off date: 29 September 2020. The study is ongoing.
Pre-assignment Details: Participants enrolled in single arm in this study to receive brigatinib 90/180 mg. The first 9 participants were assessed for initial safety in 'Safety Evaluation Lead-in Part'. Once safety was confirmed, participants were further enrolled in same arm. Data for outcome measures were assessed based on treatment taken before screening: Main Cohort(at least 1 line of prior treatment); Sub-Cohort(with 2 prior ALK-TKIs treatment); TKI-Naive Expansion Cohort(no prior treatment).
Groups:
- Brigatinib 90 mg/180 mg: Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onwards in 28-day cycles until investigator-assessed progressive disease (PD) or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to 34 cycles till data cut-off date: 29 September 2020.
Period: Overall Study
Arm/Group | Brigatinib 90 mg/180 mg
Started | 104
Safety Evaluation Lead-in Part (Safety Evaluation Lead-in Part included participants with or without prior ALK-TKI treatment. Although the protocol allowed both refractory and TKI-naive participants to enroll in the Safety Evaluation Lead-in Part, all enrolled participants had history of prior ALK-TKI and were thus included in the efficacy evaluation in All Refractory Participants Cohort.) | 9
Refractory Expansion Part: Main Cohort (Main Cohort of the Refractory Expansion Part includes participants who had previously received alectinib (as their only ALK inhibitor) or both crizotinib and alectinib.) | 47
Refractory Expansion Part: Sub-Cohort (Sub-Cohort of the Refractory Expansion Part included participants with all sequences of ALK inhibitors other than the Main Cohort, and up to 2 prior ALK inhibitor(s).) | 16
Refractory Expansion Part (Refractory Expansion Part included participants from the Main Cohort and Sub-Cohort.) | 63
All Refractory Participants (All Refractory Participants included all participants from the Main Cohort and Sub-Cohort of the Refractory Expansion Part, and Safety Evaluation Lead-in Part.) | 72
TKI-Naive Expansion Cohort (TKI-Naive Expansion Cohort included participants with no prior ALK-TKI treatment.) | 32
Completed (Completed = Participants who completed the treatment.) | 0
Completed | 0
Not Completed | 104
Not completed — Ongoing | 41
Not completed — Adverse Event | 4
Not completed — Progressive Disease | 58
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included participants who received at least 1 dose of study drug.
Groups:
- Brigatinib 90 mg/180 mg: Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onwards in 28-day cycles until investigator-assessed PD or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to 34 cycles till data cut-off date: 29 September 2020.
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 104

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) in the Main Cohort of the Refractory Expansion Part
Description: Confirmed ORR: Percentage of participants confirmed to have achieved complete response(CR) or partial response(PR) per Independent Review Committee(IRC) using Response Evaluation Criteria in Solid Tumors(RECIST) version 1.1 after the initiation of study treatment(confirmed ≥4 weeks after initial response). CR(target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR(non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size(<10 mm short axis) and normalization of tumor marker level. PR(target lesions): at least 30% decrease in sum of the longest diameters(SLD) of target lesions, taking as reference Baseline sum diameters. As pre-specified in the protocol, this outcome measure was assessed and reported data only in the participants with at least 1 line of prior treatment(called as Main Cohort) of the Refractory Expansion Part.
Time Frame: From the start of study treatment up to confirmed CR or PR (Up to approximately 23 months)
Population: Full Analysis Set-P (FAS-P) Population is a subset of the Full Analysis Set (FAS) Population and included first 47 participants in the Main Cohort of the Refractory Expansion Part.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Refractory Expansion Part: Main Cohort: Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onwards in 28-day cycles until investigator-assessed PD or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to 31 cycles till data cut-off date: 29 September 2020. Participants who had previously received only alectinib or both alectinib and crizotinib formed a part of the Main Cohort of the Refractory Expansion Part.
Arm/Group | Refractory Expansion Part: Main Cohort
Number analyzed (Participants) | 47
percentage of participants | 34.0 [20.864 to 49.313]

2. Primary Outcome: 12 Months Progression-Free Survival (PFS) Rate in the Tyrosine Kinase Inhibitor (TKI) Naïve Expansion Cohort
Description: 12 months PFS rate was defined as the percentage of the participants who did not have PFS events (PD per IRC using RECIST version 1.1, or death by any cause) at 12 months after the start of study treatment. PD for target lesion: SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm. PD for non-target lesion: unequivocal progression of existing nontarget lesions. Kaplan-Meier method was used for analysis of percentage of participants who achieved PFS of 12 months. As pre-specified in the protocol, this outcome measure was assessed and reported data only in the TKI-Naïve Expansion Cohort (participants with no prior treatment).
Time Frame: From the start of study treatment up to Month 12
Population: Participants from the FAS Population who received at least 1 dose of study drug in the TKI-Naïve Expansion Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TKI-Naive Expansion Cohort: Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onwards in 28-day cycles until investigator-assessed PD or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to 22 cycles till data cut-off date: 29 September 2020. Participants who had not received any prior TKIs including ALK-TKIs formed a part of the TKI-Naive Expansion Cohort.
Arm/Group | TKI-Naive Expansion Cohort
Number analyzed (Participants) | 32
percentage of participants | 93.0 [79.20 to 97.75]

3. Secondary Outcome: Confirmed ORR as Assessed by an IRC in All Refractory Participants and TKI-Naïve Expansion Cohort
Description: Confirmed ORR was defined as percentage of participants who were confirmed to have achieved CR or PR per an IRC using RECIST version 1.1 after initiation of study treatment (confirmed ≥4 weeks after initial response). CR for target lesion response: disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion response: disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in SLD of target lesions, taking as reference baseline sum diameters. As pre-specified in the protocol, the data for this outcome measure is reported based on previous treatment as: All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the start of study treatment up to confirmed CR or PR till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. Number analyzed are the number of participants in each cohort. Data is reported per cohort, based on the previous treatment: All Refractory Participants including Main Cohort, Sub-cohort and Safety Lead-in Cohort and and no treatment: TKI-Naive Expansion Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
percentage of participants
  All Refractory Participants: number analyzed (Participants) | 72
  All Refractory Participants | 31.9 [21.442 to 43.986]
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | 96.9 [83.783 to 99.921]

4. Secondary Outcome: Confirmed ORR as Assessed by the Investigator in Main Cohort of the Refractory Expansion Part, Safety Evaluation Lead-in Part, and TKI-Naive Expansion Cohort
Description: Confirmed ORR was defined as the percentage of the participants who were confirmed to have achieved CR or PR per the investigator using RECIST version 1.1 after the initiation of study treatment (confirmed ≥4 weeks after initial response). CR for target lesion response: disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion response: disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part and TKI-Naive Expansion Cohort. The Safety Evaluation Lead-in Part was excluded from the analysis.
Time Frame: as for outcome 3
Population: Main Cohort of Refractory Expansion Part and TKI-Naive Expansion Cohort participants from FAS, included all participants who received at least one dose of the study drug. Number analyzed are the number of participants analyzed for each cohort. Data is reported for per cohort separately: Main Cohort of Refractory Expansion Part and TKI-Naive Expansion Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 79
percentage of participants
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | 38.3 [24.507 to 53.620]
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | 93.8 [79.193 to 99.234]

5. Secondary Outcome: Duration of Response (DOR) as Assessed by an IRC in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: DOR was assessed by an IRC, per RECIST version 1.1. DOR was defined as the time between the first documentation of objective tumor response (CR or PR) and the first subsequent documentation of objective PD or death due to any cause, whichever occurs first. PD for target lesion: SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm. PD for non-target lesion: unequivocal progression of existing nontarget lesions. Only responders were analyzed for this outcome measure. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From first dose at 8-week intervals through Cycle 15 (each cycle=28 days) and at 12-week intervals thereafter until disease progression or death, whichever occurs first till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. Only responders were analyzed for this outcome measure. Number analyzed are the number of responder population in each cohort. Data is reported for each cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 54
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 16
  Main Cohort of Refractory Expansion Participants | 11.8 [5.5 to 16.4]
  All Refractory Participants: number analyzed (Participants) | 23
  All Refractory Participants | 16.4 [5.6 to NA] — Upper limit of 95% confidence interval (CI) was not reached due to low number of responders with events.
  TKI-Naive Participants: number analyzed (Participants) | 31
  TKI-Naive Participants | NA [13.9 to NA] — Median and upper limit of 95% CI were not reached due to low number of responders with events.

6. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by an IRC in the Main Cohort of the Refractory Expansion Part, and All Refractory Participants
Description: PFS was assessed by an IRC, per RECIST version 1.1. PFS was defined as the time from the start of study treatment to the first documentation of objective PD or to death due to any cause, whichever occurs first. PD for target lesion: SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm. PD for non-target lesion: unequivocal progression of existing nontarget lesions. This outcome measure reports the data in refractory participants only and data is reported per cohort separately for Main Cohort of the Refractory Expansion Part, and for All Refractory Participants.
Time Frame: From the start of the treatment up to disease progression or death due to any cause, whichever comes first till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: Refractory participants from the FAS population, including participants who received at least one dose of the study drug had a history of prior ALK-TKI treatment to which they were refractory. FAS-P Population=subset of the FAS Population and included first 47 participants in the Main Cohort of the Refractory Expansion Part. Number analyzed=number of participants in each cohort. Data is reported for each cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 72
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | 7.3 [3.7 to 9.3]
  All Refractory Participants | 7.5 [5.5 to 9.3]

7. Secondary Outcome: PFS as Assessed by an IRC in the TKI-Naive Expansion Cohort
Description: PFS was assessed by an IRC, per RECIST version 1.1. PFS was defined as the time from the start of study treatment to the first documentation of objective PD or to death due to any cause, whichever occurs first. PD for target lesion: SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest), the SLD must also demonstrate an absolute increase of at least 5 mm. PD for non-target lesion: unequivocal progression of existing nontarget lesions. This outcome measure reports data only in the TKI-Naive Expansion Cohort.
Time Frame: as for outcome 6
Population: Participants from the FAS Population who received at least 1 dose of study drug in the TKI-Naïve Expansion Cohort. Data is reported only for TKI-Naive Expansion Cohort in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI-Naive Expansion Cohort
Number analyzed (Participants) | 32
months | NA [15.7 to NA] — Median and upper limit of 90% CI were not reached due to low number of participants with events.

8. Secondary Outcome: Disease Control Rate (DCR) as Assessed by an IRC in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: DCR was assessed by an IRC, per RECIST version 1.1. DCR: percentage of participants confirmed to have achieved CR or PR or have best overall response of stable disease (SD), for 6 weeks or more after initiation of study drug. CR (target lesion): disappearance of all target lesions. CR (non-target lesions): the nontarget lesion(s) has fully resolved. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. SD (target lesion): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD (target lesion): SLD increased by at least 20% from the smallest value on study, the SLD must also demonstrate an absolute increase of at least 5 mm. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the start of the treatment up to confirmed CR or PR or SD till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. Number analyzed are the number of participants analyzed in each cohort. Data is reported per cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
percentage of participants
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | 78.7 [64.336 to 89.297]
  All Refractory Participants: number analyzed (Participants) | 72
  All Refractory Participants | 73.6 [61.897 to 83.305]
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | 96.9 [83.783 to 99.921]

9. Secondary Outcome: Time to Response as Assessed by an IRC in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: Time to response was assessed by an IRC, per RECIST version 1.1. and was defined as the time interval from the date of the first dose of study treatment until the initial observation of CR or PR for participants with confirmed CR/PR. CR(target lesion response):disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR(non-target lesion response):disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the start of the treatment up to confirmed CR or PR till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. Only responders were analyzed for this outcome measure. Number analyzed are responder population in each cohort. Data is reported for each cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Median (Full Range); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 54
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 16
  Main Cohort of Refractory Expansion Participants | 1.922 [1.25 to 9.23]
  All Refractory Participants: number analyzed (Participants) | 23
  All Refractory Participants | 1.873 [1.25 to 9.23]
  TKI-Naive Participants: number analyzed (Participants) | 31
  TKI-Naive Participants | 1.840 [0.95 to 12.88]

10. Secondary Outcome: Overall Survival (OS) as Assessed by an IRC in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the start of the treatment up to death due to any cause till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. FAS-P Population is a subset of the FAS Population and included first 47 participants in the Main Cohort of the Refractory Expansion Part. Number analyzed are the number of participants analyzed in each cohort. Data is reported per cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants including Safety Lead-in Cohort; TKI-Naive Expansion Cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | NA [14.8 to NA] — Median and upper limit of 95% CI were not reached due to low number of participants with events.
  All Refractory Participants: number analyzed (Participants) | 72
  All Refractory Participants | NA [21.7 to NA] — Median and upper limit of 95% CI were not reached due to low number of participants with events.
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | NA [NA to NA] — Median, lower and upper limit of 95% CI were not reached due to low number of participants with events.

11. Secondary Outcome: Intracranial Objective Response Rate (iORR) in Participants With Measurable Central Nervous System (CNS) Metastases at Baseline in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: Confirmed iORR was defined as the percentage of the participants who had achieved confirmed CR or PR in the intracranial CNS per modified RECIST version 1.1 as evaluated by an IRC after the initiation of study treatment. CR for target lesion: disappearance of all target lesions. CR for non-target lesions: the nontarget lesion(s) has fully resolved. PR for target lesion: at least a 30% decrease in SLD of target lesions, taking as reference the Baseline SLD. Additionally, progression of target lesions must not be present. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: as for outcome 9
Population: Participants from FAS, included all participants who received at least one dose of the study drug, with measurable CNS metastases at Baseline. FAS-P Population is a subset of the FAS Population and included first 47 participants in the Main Cohort of the Refractory Expansion Part. Number analyzed are the number of participants analyzed for each cohort. Data is reported per cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 19
percentage of participants
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 8
  Main Cohort of Refractory Expansion Participants | 25.0 [3.185 to 65.086]
  All Refractory Participants: number analyzed (Participants) | 14
  All Refractory Participants | 21.4 [4.658 to 50.798]
  TKI-Naive Participants: number analyzed (Participants) | 5
  TKI-Naive Participants | 40.0 [5.274 to 85.337]

12. Secondary Outcome: Duration of Intracranial Response (iDOR) in Participants With Measurable CNS Metastases at Baseline in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-naive Expansion Cohort
Description: iDOR was assessed by an IRC, per modified RECIST version 1.1 and was defined as the time between first documentation of objective intracranial tumor response (CR or PR) and first subsequent documentation of objective intracranial PD or death due to any cause. Participants who had systemic PD without intracranial PD were censored. CR (target lesion): disappearance of all target lesions. CR (non-target lesions):the nontarget lesion(s) has fully resolved. PR (target lesion):at least a 30% decrease in SLD of target lesions, taking as reference Baseline SLD. Progression of target lesions must not be present. CNS PD (target lesions):at least a 20% increase in SLD of target lesions, taking as reference the nadir SLD (or the baseline) and SLD must also demonstrate an absolute increase of ≥5 mm. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From first dose at 8-week intervals through Cycle 15 (each cycle=28 days) and at 12-week intervals thereafter until intracranial disease progression or death due to any cause till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: Participants from FAS, included all participants who received at least one dose of the study drug, with measurable metastases at Baseline. Data was analyzed only for the responder population. Number analyzed are responder population in each cohort. Data is reported per cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 5
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 2
  Main Cohort of Refractory Expansion Participants | 4.6 [3.7 to 5.4]
  All Refractory Participants: number analyzed (Participants) | 3
  All Refractory Participants | 5.4 [3.7 to NA] — Upper limit of 95% CI was not reached due to low number of participants with events.
  TKI-Naive Participants: number analyzed (Participants) | 2
  TKI-Naive Participants | 9.7 [5.6 to 13.8]

13. Secondary Outcome: Intracranial Progression-free Survival (iPFS) in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: iPFS was assessed by an IRC, per modified RECIST version 1.1 and was defined as the time from the start of study treatment to the first documentation of objective intracranial PD or death due to any cause, whichever occurred first. The participant who had systemic PD and withdrawn from study without intracranial PD was censored. CNS PD for target lesions: at least a 20% increase in the SLD of target lesions, taking as reference the nadir SLD (or the baseline, if the baseline is the nadir value) and the SLD must also demonstrate an absolute increase of ≥5 mm. PD for non-target lesions: the nontarget site of disease has shown unequivocal progression. As pre-specified in the protocol, this outcome measure was assessed and reports data per cohort in all participants with measurable or not measurable intracranial metastases at Baseline: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the start of the treatment up to intracranial disease progression or death due to any cause, whichever comes first till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: FAS included all participants who received at least one dose of the study drug. FAS-P Population is a subset of the FAS Population and included first 47 participants in the Main Cohort of the Refractory Expansion Part. Number analyzed are the number of participants analyzed for each cohort. Data is reported for each cohort separately: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | NA [9.2 to NA] — Median and upper limit of 95% CI were not reached due to low number of participants with events.
  All Refractory Participants: number analyzed (Participants) | 72
  All Refractory Participants | NA [15.5 to NA] — Median and upper limit of 95% CI were not reached due to low number of participants with events.
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | NA [15.7 to NA] — Median and upper limit of 95% CI were not reached due to low number of participants with events.

14. Secondary Outcome: Time on Treatment in the Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort
Description: Time on treatment was defined as the time interval from the first dose to the last dose of brigatinib. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort: Main Cohort of the Refractory Expansion Part, All Refractory Participants, and TKI-Naive Expansion Cohort.
Time Frame: From the first dose up to last dose of study drug till data cut-off date: 29 September 2020 (Up to approximately 32 months)
Population: All Refractory Participants, TKI-Naive Participants: Safety Population included all participants who received at least 1 dose of study drug. Main Cohort of Refractory Expansion: FAS-P Population is a subset of FAS including first 47 participants in the Main Cohort of the Refractory Expansion Part. Number analyzed = participants in each cohort: Main Cohort of Refractory Expansion Part; All Refractory Participants; TKI-Naive Expansion Cohort.
Measure: Median (Full Range); unit: months
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 104
months
  Main Cohort of Refractory Expansion Participants: number analyzed (Participants) | 47
  Main Cohort of Refractory Expansion Participants | 7.50 [0.2 to 20.0]
  All Refractory Participants: number analyzed (Participants) | 72
  All Refractory Participants | 8.20 [0.2 to 22.4]
  TKI-Naive Participants: number analyzed (Participants) | 32
  TKI-Naive Participants | 13.80 [0.4 to 19.3]

15. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes (PROs) of Health-Related Quality of Life (HRQOL) Scores and Symptoms as Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQC30) Subscale Score
Description: EORTC QLQ-C30 contains 30 items - 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a QOL scale. Out of 30, 28 questions had 4 response levels (not at all, a little, quite a bit, and very much); 2 questions for global health status had score of 1 to 7 (very poor to excellent) to evaluate overall health and QOL. Each subscale raw score including global health status was transformed to a total score of 0 to 100. For functional scales, global health status scale, higher scores=better QOL (positive change from Baseline=improvement). For symptom scales, lower scores=better QOL (negative change from Baseline=improvement). As pre-specified in protocol, this outcome measure was assessed and reports data per cohort: Refractory Expansion Participants (including Main Cohort and Sub-Cohort), and TKI-Naive Expansion Cohort.
Time Frame: Refractory Expansion Participants: Baseline and Cycle 22 - each cycle was of 28 days; TKI-Naive Participants: Baseline and Cycle 19 - each cycle was of 28 days
Population: Refractory Expansion Part and TKI-Naive Expansion Cohort participants from FAS, included all participants who received at least one dose of the study drug. Number analyzed are participants analyzed in each cohort for the specific category at the given timepoint. Data is reported for each cohort separately: Refractory Expansion Part; TKI-Naive Expansion Cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 95
score on a scale
  Refractory Expansion Participants (Global Health Status): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Global Health Status): Baseline | 64.3 (24.17)
  Refractory Expansion Participants (Global Health Status): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Global Health Status): Change from Baseline at Cycle 22 | -12.8 (38.92)
  Refractory Expansion Participants (Physical Functioning): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Physical Functioning): Baseline | 88.7 (16.98)
  Refractory Expansion Participants (Physical Functioning): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Physical Functioning): Change From Baseline at Cycle 22 | 1.8 (3.50)
  Refractory Expansion Participants (Role Functioning): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Role Functioning): Baseline | 85.5 (21.22)
  Refractory Expansion Participants (Role Functioning): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Role Functioning): Change From Baseline at Cycle 22 | 4.3 (8.50)
  Refractory Expansion Participants (Emotional Functioning): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Emotional Functioning): Baseline | 87.5 (15.53)
  Refractory Expansion Participants (Emotional Functioning): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Emotional Functioning): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Cognitive Functioning): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Cognitive Functioning): Baseline | 87.8 (16.72)
  Refractory Expansion Participants (Cognitive Functioning): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Cognitive Functioning): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Social Functioning): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Social Functioning): Baseline | 86.8 (20.97)
  Refractory Expansion Participants (Social Functioning): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Social Functioning): Change From Baseline at Cycle 22 | 4.3 (8.50)
  Refractory Expansion Participants (Fatigue): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Fatigue): Baseline | 22.3 (22.73)
  Refractory Expansion Participants (Fatigue): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Fatigue): Change from Baseline at Cycle 22 | 5.5 (11.00)
  Refractory Expansion Participants (Nausea and Vomiting): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Nausea and Vomiting): Baseline | 4.5 (14.16)
  Refractory Expansion Participants (Nausea and Vomiting): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Nausea and Vomiting): Change from Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Pain): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Pain): Baseline | 15.3 (17.46)
  Refractory Expansion Participants (Pain): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Pain): Change from Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Dyspnoea): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Dyspnoea): Baseline | 20.6 (25.73)
  Refractory Expansion Participants (Dyspnoea): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Dyspnoea): Change from Baseline at Cycle 22 | -8.3 (16.50)
  Refractory Expansion Participants (Insomnia): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Insomnia): Baseline | 17.9 (21.41)
  Refractory Expansion Participants (Insomnia): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Insomnia): Change from Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Appetite loss): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Appetite loss): Baseline | 13.2 (25.75)
  Refractory Expansion Participants (Appetite loss): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Appetite loss): Change from Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Constipation): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Constipation): Baseline | 14.2 (22.94)
  Refractory Expansion Participants (Constipation): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Constipation): Change from Baseline at Cycle 22 | 8.3 (16.50)
  Refractory Expansion Participants (Diarrhoea): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Diarrhoea): Baseline | 5.3 (14.90)
  Refractory Expansion Participants (Diarrhoea): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Diarrhoea): Change from Baseline at Cycle 22 | 24.8 (16.50)
  Refractory Expansion Participants (Financial Difficulties): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Financial Difficulties): Baseline | 14.7 (24.49)
  Refractory Expansion Participants (Financial Difficulties): Change from Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Financial Difficulties): Change from Baseline at Cycle 22 | 0.0 (0.00)
  TKI-Naive Participants (Global Health Status): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Global Health Status): Baseline | 64.8 (23.15)
  TKI-Naive Participants (Global Health Status):Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Global Health Status):Change from Baseline at Cycle 19 | 1.3 (13.32)
  TKI-Naive Participants (Physical Functioning): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Physical Functioning): Baseline | 88.1 (12.10)
  TKI-Naive Participants (Physical Functioning): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Physical Functioning): Change from Baseline at Cycle 19 | -6.5 (12.86)
  TKI-Naive Participants (Role Functioning): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Role Functioning): Baseline | 81.3 (21.89)
  TKI-Naive Participants (Role Functioning): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Role Functioning): Change From Baseline at Cycle 19 | -11.0 (17.04)
  TKI-Naive Participants (Emotional Functioning): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Emotional Functioning): Baseline | 80.5 (14.14)
  TKI-Naive Participants (Emotional Functioning): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Emotional Functioning): Change From Baseline at Cycle 19 | 6.8 (9.72)
  TKI-Naive Participants (Cognitive Functioning): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Cognitive Functioning): Baseline | 88.5 (16.09)
  TKI-Naive Participants (Cognitive Functioning): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Cognitive Functioning): Change From Baseline at Cycle 19 | -2.7 (16.34)
  TKI-Naive Participants (Social Functioning): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Social Functioning): Baseline | 77.1 (23.50)
  TKI-Naive Participants (Social Functioning): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Social Functioning): Change From Baseline at Cycle 19 | 0.2 (21.19)
  TKI-Naive Participants (Fatigue): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Fatigue): Baseline | 23.4 (18.34)
  TKI-Naive Participants (Fatigue): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Fatigue): Change From Baseline at Cycle 19 | 3.7 (11.36)
  TKI-Naive Participants (Nausea and Vomiting): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Nausea and Vomiting): Baseline | 1.6 (5.03)
  TKI-Naive Participants (Nausea and Vomiting): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Nausea and Vomiting): Change From Baseline at Cycle 19 | 2.8 (6.94)
  TKI-Naive Participants (Pain): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Pain): Baseline | 22.9 (23.04)
  TKI-Naive Participants (Pain): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Pain): Change from Baseline at Cycle 19 | 2.7 (12.04)
  TKI-Naive Participants (Dyspnoea): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Dyspnoea): Baseline | 20.7 (21.98)
  TKI-Naive Participants (Dyspnoea): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Dyspnoea): Change from Baseline at Cycle 19 | -0.2 (29.74)
  TKI-Naive Participants (Insomnia): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Insomnia): Baseline | 21.7 (21.67)
  TKI-Naive Participants (Insomnia): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Insomnia): Change from Baseline at Cycle 19 | -10.8 (27.27)
  TKI-Naive Participants (Appetite loss): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Appetite loss): Baseline | 13.5 (20.46)
  TKI-Naive Participants (Appetite loss): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Appetite loss): Change from Baseline at Cycle 19 | -11.0 (26.94)
  TKI-Naive Participants (Constipation): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Constipation): Baseline | 9.3 (17.35)
  TKI-Naive Participants (Constipation): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Constipation): Change from Baseline at Cycle 19 | -5.5 (13.47)
  TKI-Naive Participants (Diarrhoea): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Diarrhoea): Baseline | 4.1 (11.09)
  TKI-Naive Participants (Diarrhoea): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Diarrhoea): Change from Baseline at Cycle 19 | 5.5 (24.84)
  TKI-Naive Participants (Financial Difficulties): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Financial Difficulties): Baseline | 20.7 (21.98)
  TKI-Naive Participants (Financial Difficulties): Change from Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Financial Difficulties): Change from Baseline at Cycle 19 | -11.0 (17.04)

16. Secondary Outcome: Change From Baseline in HRQOL Scores and Symptoms of Lung Cancer as Assessed With the EORTC QLQ- Lung Cancer (LC) 13 (QLQ-LC13) Subscale Score
Description: HRQOL scores was assessed with EORTC, its lung cancer module QLQ-LC13. QLQ-LC13 contains 13 questions (4-point scale where 1=Not at all [best] to 4=Very much [worst]) assessing lung cancer-associated symptoms [cough, hemoptysis, dyspnea, and site-specific pain (chest, arm or shoulder, other parts)], treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Subscale score range: 0 to 100. Higher symptom score = greater degree of symptom severity. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort only in the Refractory Expansion Participants (including Main Cohort and Sub-cohort), and TKI-Naive Expansion Cohort.
Time Frame: as for outcome 15
Population: FAS included all participants who received at least one dose of the study drug. Number analyzed are participants analyzed in each cohort for the specific category at the given timepoint. Data is reported for each cohort separately: Refractory Expansion Part; TKI-Naive Expansion Cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 95
score on a scale
  Refractory Expansion Participants (Dyspnea): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Dyspnea): Baseline | 17.0 (18.30)
  Refractory Expansion Participants (Dyspnea):Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Dyspnea):Change From Baseline at Cycle 22 | -2.8 (5.50)
  Refractory Expansion Participants (Coughing): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Coughing): Baseline | 32.7 (29.70)
  Refractory Expansion Participants (Coughing): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Coughing): Change From Baseline at Cycle 22 | 0.3 (47.14)
  Refractory Expansion Participants (Haemoptysis): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Haemoptysis): Baseline | 5.3 (16.01)
  Refractory Expansion Participants (Haemoptysis): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Haemoptysis): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Sore Mouth): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Sore Mouth): Baseline | 2.1 (8.11)
  Refractory Expansion Participants (Sore Mouth): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Sore Mouth): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Dysphagia): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Dysphagia): Baseline | 3.1 (9.76)
  Refractory Expansion Participants (Dysphagia): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Dysphagia): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Peripheral Neuropathy): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Peripheral Neuropathy): Baseline | 4.2 (12.64)
  Refractory Expansion Participants (Peripheral Neuropathy): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Peripheral Neuropathy): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Alopecia): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Alopecia): Baseline | 4.7 (16.76)
  Refractory Expansion Participants (Alopecia): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Alopecia): Change From Baseline at Cycle 22 | 0.0 (0.00)
  Refractory Expansion Participants (Pain in Chest): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Pain in Chest): Baseline | 12.1 (19.16)
  Refractory Expansion Participants (Pain in Chest): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Pain in Chest): Change From Baseline at Cycle 22 | -8.3 (16.50)
  Refractory Expansion Participants (Pain in Arm or Shoulder): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Pain in Arm or Shoulder): Baseline | 10.5 (18.72)
  Refractory Expansion Participants (Pain in Arm or Shoulder): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Pain in Arm or Shoulder): Change From Baseline at Cycle 22 | 8.3 (16.50)
  Refractory Expansion Participants (Pain in Other Parts): Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants (Pain in Other Parts): Baseline | 11.0 (16.82)
  Refractory Expansion Participants (Pain in Other Parts): Change From Baseline at Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants (Pain in Other Parts): Change From Baseline at Cycle 22 | 0.0 (0.00)
  TKI-Naive Participants (Dyspnea): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Dyspnea): Baseline | 16.5 (17.52)
  TKI-Naive Participants (Dyspnea): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Dyspnea): Change From Baseline at Cycle 19 | 7.3 (17.96)
  TKI-Naive Participants (Coughing): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Coughing): Baseline | 36.3 (29.84)
  TKI-Naive Participants (Coughing): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Coughing): Change From Baseline at Cycle 19 | -11.2 (17.30)
  TKI-Naive Participants (Haemoptysis): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Haemoptysis): Baseline | 3.1 (9.77)
  TKI-Naive Participants (Haemoptysis): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Haemoptysis): Change From Baseline at Cycle 19 | -5.5 (13.47)
  TKI-Naive Participants (Sore Mouth): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Sore Mouth): Baseline | 8.3 (16.88)
  TKI-Naive Participants (Sore Mouth): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Sore Mouth): Change From Baseline at Cycle 19 | 0.0 (20.87)
  TKI-Naive Participants (Dysphagia): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Dysphagia): Baseline | 7.3 (16.32)
  TKI-Naive Participants (Dysphagia): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Dysphagia): Change From Baseline at Cycle 19 | -5.5 (24.84)
  TKI-Naive Participants (Peripheral Neuropathy): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Peripheral Neuropathy): Baseline | 8.3 (22.39)
  TKI-Naive Participant (Peripheral Neuropathy): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participant (Peripheral Neuropathy): Change From Baseline at Cycle 19 | 0.0 (20.87)
  TKI-Naive Participants (Alopecia): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Alopecia): Baseline | 3.1 (9.77)
  TKI-Naive Participants (Alopecia): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Alopecia): Change From Baseline at Cycle 19 | 0.0 (20.87)
  TKI-Naive Participants (Pain in Chest): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Pain in Chest): Baseline | 13.4 (16.47)
  TKI-Naive Participants (Pain in Chest): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Pain in Chest): Change From Baseline at Cycle 19 | -11.0 (17.04)
  TKI-Naive Participants (Pain in Arm or Shoulder): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Pain in Arm or Shoulder): Baseline | 15.5 (23.87)
  TKI-Naive Participants (Pain in Arm or Shoulder): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Pain in Arm or Shoulder): Change From Baseline at Cycle 19 | -5.5 (24.84)
  TKI-Naive Participants (Pain in Other Parts): Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants (Pain in Other Parts): Baseline | 19.7 (20.44)
  TKI-Naive Participants (Pain in Other Parts): Change From Baseline at Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants (Pain in Other Parts): Change From Baseline at Cycle 19 | 5.5 (13.47)

17. Secondary Outcome: Number of Participants With Responses to HRQOL Scores and Symptoms of Lung Cancer as Assessed With the EuroQol 5-Dimensional Questionnaire (EQ-5D-5L) Score
Description: EQ-5D-5L comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, 5= extremely severe problems. Higher scores indicated greater levels of problems across the five dimensions. As pre-specified in the protocol, this outcome measure assessed and reports data per cohort only in the Refractory Expansion Participants (including Main Cohort and Sub-cohort), and TKI-Naive Expansion Cohort. Number of participants with a particular score at the given timepoint is reported. Only categories with data are reported.
Time Frame: Refractory Expansion Participants: Cycle 22 - each cycle was of 28 days; TKI-Naive Participants: Cycle 19 - each cycle was of 28 days
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 95
Participants
  Refractory Expansion Participants(Score=1, Mobility: Have no problems walking): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=1, Mobility: Have no problems walking) | 4
  Refractory Expansion Participants(Score=1, Selfcare: Have no problems washing/dressing myself): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=1, Selfcare: Have no problems washing/dressing myself) | 4
  Refractory Expansion Participants(Score=1, Activity: Have no problems doing usual activities): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=1, Activity: Have no problems doing usual activities) | 4
  Refractory Expansion Participants(Score=1, Pain: Have no pain or discomfort): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=1, Pain: Have no pain or discomfort) | 3
  Refractory Expansion Participants(Score=2, Pain: Have slight pain or discomfort): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=2, Pain: Have slight pain or discomfort) | 1
  Refractory Expansion Participants(Score=1, Anxiety: Not anxious or depressed): number analyzed (Participants) | 4
  Refractory Expansion Participants(Score=1, Anxiety: Not anxious or depressed) | 4
  TKI-Naive Participants(Score=1, Mobility: Have no problems walking): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=1, Mobility: Have no problems walking) | 4
  TKI-Naive Participants(Score=2, Mobility: Have slight problems walking): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=2, Mobility: Have slight problems walking) | 2
  TKI-Naive Participants(Score=1, Selfcare: Have no problems washing/dressing myself): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=1, Selfcare: Have no problems washing/dressing myself) | 6
  TKI-Naive Participants(Score=1, Activity: Have no problems doing my usual activities): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=1, Activity: Have no problems doing my usual activities) | 6
  TKI-Naive Participants(Score=1, Pain: Have no pain or discomfort): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=1, Pain: Have no pain or discomfort) | 1
  TKI-Naive Participants(Score=2, Pain: Have slight pain or discomfort): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=2, Pain: Have slight pain or discomfort) | 5
  TKI-Naive Participants(Score=1, Anxiety: Not anxious or depressed): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=1, Anxiety: Not anxious or depressed) | 4
  TKI-Naive Participants(Score=2,Anxiety: Slightly anxious or depressed): number analyzed (Participants) | 6
  TKI-Naive Participants(Score=2,Anxiety: Slightly anxious or depressed) | 2

18. Secondary Outcome: Change From Baseline in HRQOL Scores and Symptoms of Lung Cancer as Assessed With the EuroQol Visual Analogue Scale (EQ VAS) Score
Description: The EQ VAS records the respondent's self-rated health on a 20 centimeter (cm), vertical, visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). As pre-specified in the protocol, this outcome measure assessed and reports data per cohort only in the Refractory Expansion Participants (including Main Cohort and Sub-cohort), and TKI-Naive Expansion Cohort.
Time Frame: as for outcome 15
Population: FAS included all participants who received at least one dose of the study drug. Number analyzed are participants analyzed in each cohort at the given timepoint. Data is reported for each cohort separately: Refractory Expansion Part; TKI-Naive Expansion Cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brigatinib 90 mg/180 mg
Number analyzed (Participants) | 95
score on a scale
  Refractory Expansion Participants: Baseline: number analyzed (Participants) | 63
  Refractory Expansion Participants: Baseline | 72.0 (19.65)
  Refractory Expansion Participants: Change from Baseline to Cycle 22: number analyzed (Participants) | 4
  Refractory Expansion Participants: Change from Baseline to Cycle 22 | 4.3 (11.93)
  TKI-Naive Participants: Baseline: number analyzed (Participants) | 32
  TKI-Naive Participants: Baseline | 73.3 (21.10)
  TKI-Naive Participants: Change from Baseline to Cycle 19: number analyzed (Participants) | 6
  TKI-Naive Participants: Change from Baseline to Cycle 19 | 3.2 (6.01)

19. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Brigatinib on Cycle 1 Days 1 and 22
Description: As pre-specified in the protocol, this outcome measure was assessed only in the participants with or without prior ALK-TKI treatment called as the Safety Evaluation Lead-in Part.
Time Frame: Pre-dose and at multiple time points (0.5, 1, 2, 4, 6, 8, 12, 24; up to 24 hrs) post-dose of Cycle 1 Days 1 and 22 (each cycle = 28 days)
Population: Pharmacokinetic (PK) Population included participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist for Safety Evaluation Lead-in Part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Safety Evaluation Lead-in Part: Brigatinib 90 mg, tablets, orally, QD for first 7 days followed by brigatinib, 180 mg, tablets, orally, QD in Cycle 1 of 28 days followed by brigatinib 180 mg, tablets, orally, QD in Cycle 2 and onwards in 28-day cycles until investigator-assessed PD or intolerable toxicity, withdrawal of consent, or discontinuation for any other reason, whichever comes first up to 34 cycles till data cut-off date: 29 September 2020. Participants with or without prior ALK-TKI treatment formed a part of the Safety Evaluation Lead-in Part.
Arm/Group | Safety Evaluation Lead-in Part
Number analyzed (Participants) | 9
ng/mL
  Cycle 1 Day 1 | 414.0 (52.2)
  Cycle 1 Day 22 | 2119 (62.5)

20. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Brigatinib on Cycle 1 Days 1 and 22
Description: as for outcome 19
Time Frame: as for outcome 19
Population: PK Population included participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist for Safety Evaluation Lead-in Part.
Measure: Median (Full Range); unit: hour
Arm/Group | Safety Evaluation Lead-in Part
Number analyzed (Participants) | 9
hour
  Cycle 1 Day 1 | 3.980 [1.02 to 7.88]
  Cycle 1 Day 22 | 2.080 [1.12 to 6.03]

21. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post-dose for Brigatinib on Cycle 1 Days 1 and 22
Description: as for outcome 19
Time Frame: as for outcome 19
Population: PK Population included participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist for Safety Evaluation Lead-in Part. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Safety Evaluation Lead-in Part
Number analyzed (Participants) | 9
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 8
  Cycle 1 Day 1 | 5045 (48.4)
  Cycle 1 Day 22 | 31130 (60.0)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug or initiation of the subsequent anticancer therapies, whichever comes first (Up to data cut-off date: 29 September 2020 [Up to approximately 32 months])
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Brigatinib 90 mg/180 mg
All-Cause Mortality (participants affected / at risk) | 21/104
Serious Adverse Events (participants affected / at risk) | 37/104
Other Adverse Events (participants affected / at risk) | 103/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90 mg/180 mg (N=104)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 4
Hepatic infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Blood insulin increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 2
Brain oedema (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Thrombophlebitis migrans (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90 mg/180 mg (N=104)
Anaemia (Blood and lymphatic system disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 47
Stomatitis (Gastrointestinal disorders) | 34
Nausea (Gastrointestinal disorders) | 33
Constipation (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 16
Pyrexia (General disorders) | 19
Malaise (General disorders) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 10
Upper respiratory tract infection (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 9
Blood creatine phosphokinase increased (Investigations) | 81
Aspartate aminotransferase increased (Investigations) | 36
Lipase increased (Investigations) | 35
Amylase increased (Investigations) | 33
Alanine aminotransferase increased (Investigations) | 24
Blood alkaline phosphatase increased (Investigations) | 15
Blood creatinine increased (Investigations) | 7
Blood lactate dehydrogenase increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 17
Peripheral sensory neuropathy (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 20
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 10
Hypertension (Vascular disorders) | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03410108/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03410108/SAP_001.pdf